CLINICAL TRIAL: NCT01743950
Title: A Phase II Study of Pulse Reduced Dose Rate Radiation Therapy With Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO11374; NCI-2012-02775 (Registry Identifier: NCI Trial ID); 2012-0648 (Other: Institutional Review Board); 2017-0683 (Other: Institutional Review Board); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison); Protocol Version 10/14/2020 (Other: UW Madison)
Record Dates: First submitted 2012-11-27; First posted 2012-12-06 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Glioma
Keywords: Glioblastoma; anaplastic glioma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Bevacizumab; Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Bevacizumab-naïve with recurrent IDH wildtype high grade glioma (Active Comparator): 27fractions over 5.5weeks of PRDR radiation with bevacizumab followed by adjuvant bevacizumab until time of progression
  Interventions: Drug: Bevacizumab; Radiation: PRDR
- Bevacizumab-exposed with refractory recurrent IDH wildtype high grade glioma (Active Comparator): 27fractions over 5.5weeks of PRDR radiation with bevacizumab followed by adjuvant bevacizumab until time of progression
  Interventions: Drug: Bevacizumab; Radiation: PRDR
- Bevacizumab-naïve with recurrent IDH mutant glioma (Active Comparator): 27fractions over 5.5weeks of PRDR radiation with bevacizumab followed by adjuvant bevacizumab until time of progression
  Interventions: Drug: Bevacizumab; Radiation: PRDR
- Bevacizumab-exposed with recurrent IDH mutant glioma (Active Comparator): 27fractions over 5.5weeks of PRDR radiation with bevacizumab followed by adjuvant bevacizumab until time of progression
  Interventions: Drug: Bevacizumab; Radiation: PRDR

INTERVENTIONS:
Drug: Bevacizumab — 10mg/kg every 2weeks.
Radiation: PRDR — Daily dose of 2.0gy delivered in .2gy pulses for a total of 54gy over 5.5 weeks and 27 fractions. In the rare instance of the presence of extensive disease requiring essentially whole brain radiation, a total daily dose of 1.8 Gy delivered in .2 Gy pulses for 23 fractions to a total dose of 41.4 Gy will be utilized.
  Other Names: re-irradiation

SUMMARY:
To determine the efficacy of Pulse Reduced Dose Rate (PRDR) radiation when given in 27 fraction over 5.5 weeks with concurrent bevacizumab followed by adjuvant bevacizumab until time of progression in patients with recurrent high grade gliomas (grade III and grade IV). Patients will be placed in 1 of 4 groups based on their histologic diagnosis and prior exposure to bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or molecularly confirmed Grade 3 or 4 glioma, IDH mutant or wildtype, as defined by the 2021 WHO guidelines
* Recurrent disease based on combination of clinical, imaging or histologic confirmation
* Must have previously received radiation and temozolomide to treat their glioma
* Bevacizumab naive patients must be > 5 months post completion of initial radiation therapy
* Bevacizumab exposed patients must be > 3 months post completion of initial radiation therapy
* Age must be >18years, KPS must be greater than 60
* Hematology, chemistry and a urinalysis must meet protocol specified criteria

Exclusion Criteria:

* Pregnant or breastfeeding
* Uncontrolled hypertension (>160/90mmHg)
* Prior malignancy unless treated >1 year prior to study and have been without treatment and disease free for 1 yr
* active second malignancy unless non-melanoma skin cancer or cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Overall survival | end of study, which will be an average of 12 months
  time of first dose of PDRD+ Bevacizumab until time of death

SECONDARY OUTCOMES:
Incidence of Adverse Events | up to 30 days post last dose of bevacizumab
  time of first dose of PDRD+ Bevacizumab until time of death. All changes from baseline assessment will be recorded until 30 days post last dose of bevacizumab, assessed using the NCI CTCAE version 4.0 criteria.
Incidence of Late Toxicities | from 90 days post radiotherapy until time of death
  Late toxicity that is likely attributable to re-irradiation or bevacizumab will be recorded.
progression free survival | at 3 months for bevacizumab exposed patients, at 6 and 12 months for all patients
  Progression free survival (PFS) will be defined as the time from the first study treatment to the first occurrence of disease progression or death.
Change in Mini Mental State Exam (MMSE) Score | baseline and then approximately every 8 weeks for 18 months
  The MMSE survey is a clinician facilitated instrument scored on a scale of 0-30 where scores of 0-17 indicate severe cognitive impairment, 18-23 indicate mild cognitive impairment, and 24-30 indicate no cognitive impairment.
Change in Participant Reported FACT-BR Score | baseline and then approximately every 8 weeks for 18 months
  The Functional Assessment of Cancer Therapy - Brain (FACT-BR) instrument is a 50-item survey with each item scored on a 5 point likert scale where 0 is 'not at all' and 4 is 'very much'. The total possible range of scores is 0-200 where higher scores indicate higher quality of life.
Change in Participant Reported FACIT-F Score | baseline and then approximately every 8 weeks for 18 months
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) instrument is a 13-item survey with each item scored on a 5 point likert scale where 0 is 'not at all' and 4 is 'very much'. The total possible range of scores is from 0-52 where higher scores indicate better quality of life. A score of less than 30 indicates severe fatigue.
Change in Karnofsky Performance Status | baseline and then approximately every 8 weeks for 18 months
  The Karnofsky Performance Status measures a cancer patient's ability to perform ordinary tasks. It is score from 0-100 where 0 means a person has died, less than 40 is various degrees of unable to care for oneself, 50-70 is unable to work but can care for personal needs with variable assistance, and 80-100 is able to carry on normal activity with variable symptoms of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Howard, MD, Principal Investigator — University of Wisconsin, Madison; H. Ian Robins, MD, Ph.D, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/